CLINICAL TRIAL: NCT04805879
Title: A Clinical Trial to Evaluate the Safety and Efficacy of Fecal Microbiota Transplantation in a Population With Major Depressive Disorder
Brief Title: The Safety and Efficacy of Fecal Microbiota Transplantation in a Population With Major Depressive Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Cumming school of medicine (Unknown); The W. Garfield Westin Foundation (Unknown)
Responsible Party: Principal Investigator, Valerie Taylor, Head of Psychiatry, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB#19-0016
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Depression; Treatment Resistant Depression
Keywords: FMT; Fecal Microbiota Transplantation; Microbiome; gut brain axis; Major depression
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT capsules (Active Comparator): Each dose of FMT capsules consists of 20 capsules. The 20 over encapsulated capsules are derived from 100 grams of stool and each containing 0.67 ml of pelleted intestinal microbes.
  PArticipants will recieve a loading dose of 60 capsules over 3 consecutive days followed by a booster dose of 20 caspules 1 month after and a second similar booster dose a month after that
  Interventions: Biological: FMT oral Capsules
- Placebo oral Capsules (Placebo Comparator): Placebo casules are inactive capsules that look and weigh the same as the Active FMT caspules. Participants will follow the same schedule as the Active arm.
  Interventions: Biological: Placebo Capsules

INTERVENTIONS:
Biological: FMT oral Capsules — Each dose of FMT capsules consists of 20 capsules. The 20 over encapsulated capsules are derived from 100 grams of stool donated by a healthy indvidual that was screened to have no mental health issues or chronic or contagious doseases. Each capsule will contain 0.67 ml of pelleted intestinal microbes. Therefore it is considered that the 20 capsules are equivalent to 100 grams of stool
  Arms: FMT capsules
Biological: Placebo Capsules — Placebo Capsules that will look and weigh the same as the FMT oral capsules.
  Arms: Placebo oral Capsules

SUMMARY:
The primary goals of this proof of concept clinical trial are to determine the effectiveness, safety and tolerability of oral FMT in adults with Treatment Resistant Depression (TRD).

DETAILED DESCRIPTION:
This study is a phase 2/3, double-blinded, randomized controlled trial (RCT) in which 80 adults with TRD being treated with an approved antidepressant medication will be assigned to either FMT capsules or identically appearing placebo capsules. Participant will be followed for f for 14 weeks post FMT. This extended observation period will allow us to see, whether FMT leads to sustainable improvements in depression and changes in intestinal microbiome

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-65 years of age:

   Participants should be at least 18 years old and not older than 65 years at the day of screening
2. Have a primary diagnosis of MDD according to the M.I.N.I. International Neuropsychiatric Interview (MINI)47
3. Medical history suggestive of Treatment Resistant Depression (TRD). (inadequate response to at least 2 approved antidepressants. at least one of which is in the current episode of depression)48
4. Have been on a current treatment with a approved antidepressant at an adequate dose for at least 8 weeks
5. A MADRS score of ≥ 19 at screening and visit 2

Additional Inclusion Criteria:

- Participants who will be included in the IBS-D cohort should have a confirmed diagnosis of IBS-D as indicated by the referring gastroenterologist.

Exclusion Criteria:

* 1. Participant meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5)1 Criteria for the following conditions according to the M.I.N.I: f) Substance Use Disorder within the last 3 months. *(Criteria should include Alcohol and non-alcohol substances except Cannabis) g) Moderate or severe Substance use disorder for Cannabis use the last 3 months h) Active Anorexia Nervosa or Bulimia nervosa i) Schizophrenia or schizoaffective disorder j) Active suicidality 2. Regular intake of non-steroidal anti-inflammatory drugs, antibiotics, or iron supplements for medical purposes in the 3 months prior to study entry 3. Use of prebiotics or probiotics for medical purposes for more than 2 weeks within the last 3 months 4. Clinically diagnosed chronic gastrointestinal diseases (IBD, Crohn's disease, Ulcerative colitis, Celiac disease) 5. Conditions causing immune suppression 6. Not breastfeeding, pregnant or seeking to get pregnant during the course of this study. Be using an acceptable method of birth control (implants, injectable, combined oral contraceptives, IUDs, sexual abstinence or a vasectomized partner) 7. Reported allergy to Vancomycin or Nitazoxanide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-03-04 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Change in the MADRS total score | from baseline (pre-intervention) to the final visit (week 13)
  To evaluate the effectiveness of adjunct oral FMT as compared to placebo with currently accepted approved therapy for depression

SECONDARY OUTCOMES:
Side effects as reported on the Toronto Side Effect Scale (TSES) | from baseline (pre-intervention) to the final visit (week 13)
  The tolerability of FMT will be assessed using the Toronto Side effects Scale (TSES)
GI tolerability of patients with Irritable Bowel Syndrome (IBS) | from baseline (pre-intervention) to the final visit (week 13)
  GI tolerability will be assessed using the IBS Symptom Severity Scale (IBS SSS) and IBS specific Quality of Life (IBS-QoL) questionnaire

OTHER OUTCOMES:
To assess the effect of FMT on microbiome profile | from baseline (pre-intervention) to the final visit (week 13)
  Changes will be assessed using next generation sequencing and nuclear magnetic resonance (NMR) spectrometry
changes in inflammatory markers (Blood) | from baseline (pre-intervention) to the final visit (week 13)
  To study the changes in inflammatory markers (blood CRP)
changes in inflammatory markers (stool) | from baseline (pre-intervention) to the final visit (week 13)
  To study the changes in inflammatory markers (fecal calprotectin)
changes in serum cytokines | from baseline (pre-intervention) to the final visit (week 13)
  To study the changes in serum cytokines (IL-6, IL-10, IL-8, IFNγ and TNF)
To examine imaging changes | from baseline (pre-intervention) to the final visit (week 13)
  examine imaging changes via a structural and functional neuroimaging scan associated with FMT

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Taylor, MD, PhD, Principal Investigator — Cumming School of Medicine, University of Calgary
Locations (1):
- Cumming School of Medicine, University of Calgary, Calgary, Alberta, Canada